CLINICAL TRIAL: NCT06964074
Title: The Addition of a PEP or O-PEP Device to Nebulization With Hypertonic Saline in Patients With Cystic Fibrosis During Exacerbation
Brief Title: PEP and O-PEP Device for Nebulization in Cystic Fibrosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NITLD892510
Record Dates: First submitted 2025-03-17; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; exacerbations; chest physiotherapy; PEP device; O-PEP device
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: The physiotherapy program involves:
  Firstly, performing inhalations with hypertonic saline using one of two devices (Aerobika*OPEP with AeroEclipse XL BAN nebulizer, PARI PEP® S System with Pari LC Sprint nebulizer). The third group serves as the control group and performs inhalations using the Pari LC Sprint nebulizer. After the inhalation, participants record the amount of sputum expectorated during the inhalation and note the color of the sputum.
  Secondly, immediately after the hypertonic saline inhalation, participants use physiotherapy focused on airway clearance with the Pari O-PEP Flutter device and perform autogenic drainage for 15 breaths in one cycle. Frequency: twice a day. This cycle is repeated twice. The maximum number of cycles is five, depending on the need. Duration: 15-30 minutes. After the physiotherapy, participants also recorded the amount of expectorated secretion and noted the color of the sputum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobika with hypertonic saline nebulization (Experimental): Inhalation involves breathing through the device Aerobika with the dedicated AeroEclipse XL BAN nebulizer. The level of expiratory resistance is adjusted individually. The pressure ranges from 5 to 20 cm H2O, and the oscillation frequency is approximately 15 Hz. The inhalation duration is 10 minutes. The program duration is 10 days. The frequency is twice a day.
  Interventions: Device: Nebulization with OPEP device
- PEP with hypertonic saline nebulization (Experimental): Inhalation using the PARI PEP® S System involves breathing through the device with the dedicated Pari LC Sprint nebulizer. The level of expiratory resistance is adjusted individually. The pressure in the mid-expiratory range is 10-20 cmH2O. The inhalation duration is 10 minutes. The program duration is 10 days. The frequency is twice a day.
  Interventions: Device: Nebulization with PEP device
- hypertonic saline nebulization control group (Experimental): Inhalation with a hypertonic saline solution using a Pari LC Sprint nebulizer with a mouthpiece and nasal clip. The inhalation duration is 10 minutes. The program duration is 10 days. The frequency is twice a day..
  Interventions: Device: Nebulization with Pari LC Sprint

INTERVENTIONS:
Device: Nebulization with OPEP device — During hospitalization due to exacerbation of the bronchopulmonary disease, patients performed inhalations twice a day using one of two devices: "PARI PEP® S System" (produced by PARI, Germany) with a dedicated Pari LC Sprint nebulizer or the "Aerobika*OPEP Device" (produced by TRUDELL MEDICAL INTERNATIONAL) with a dedicated Aero Eclipse XL nebulizer, or they were in the control group where they performed inhalations in the standard way using the Pari LC Sprint nebulizer (produced by PARI, Germany). Frequency: twice daily. Inhalation duration: 10 minutes. Immediately after inhalation, each patient performed physiotherapy in the same scheme using the "Pari OPEP" device, 15 exhalations, and autogenic drainage technique according to the method's concept, with the drainage duration ranging from 15 to 30 minutes.
  Arms: Aerobika with hypertonic saline nebulization
Device: Nebulization with PEP device — During hospitalization due to exacerbation of the bronchopulmonary disease, patients performed inhalations twice a day using one of two devices: "PARI PEP® S System" (produced by PARI, Germany) with a dedicated Pari LC Sprint nebulizer or the "Aerobika*OPEP Device" (produced by TRUDELL MEDICAL INTERNATIONAL) with a dedicated Aero Eclipse XL nebulizer, or they were in the control group where they performed inhalations in the standard way using the Pari LC Sprint nebulizer (produced by PARI, Germany). Frequency: twice daily. Inhalation duration: 10 minutes. Immediately after inhalation, each patient performed physiotherapy in the same scheme using the "Pari OPEP" device, 15 exhalations, and autogenic drainage technique according to the method's concept, with the drainage duration ranging from 15 to 30 minutes.
  Arms: PEP with hypertonic saline nebulization
Device: Nebulization with Pari LC Sprint — During hospitalization due to exacerbation of the bronchopulmonary disease, patients performed inhalations twice a day using one of two devices: "PARI PEP® S System" (produced by PARI, Germany) with a dedicated Pari LC Sprint nebulizer or the "Aerobika*OPEP Device" (produced by TRUDELL MEDICAL INTERNATIONAL) with a dedicated Aero Eclipse XL nebulizer, or they were in the control group where they performed inhalations in the standard way using the Pari LC Sprint nebulizer (produced by PARI, Germany). Frequency: twice daily. Inhalation duration: 10 minutes. Immediately after inhalation, each patient performed physiotherapy in the same scheme using the "Pari OPEP" device, 15 exhalations, and autogenic drainage technique according to the method's concept, with the drainage duration ranging from 15 to 30 minutes.
  Arms: hypertonic saline nebulization control group

SUMMARY:
Physiotherapy is an essential element in the comprehensive treatment of patients with cystic fibrosis. In symptomatic individuals, from a respiratory system perspective, it should be performed regularly, as it directly contributes to slowing disease progression. Even though patients perform airway-clearing physical therapy daily, it should be intensified during exacerbations. Although solutions for effectively clearing the airways have been sought for many years, there is still no leading technique for removing secretions from the respiratory tract. Modifications during inhalation aimed at thinning and loosening the accumulated thick mucus can facilitate the effective mobilization and expectoration of secretions, thus improving patients' quality of life.

DETAILED DESCRIPTION:
The study aims to determine whether the addition of devices with positive expiratory pressure (Pari PEP System S) or positive pressure with oscillation (Aerobika) assists with hypertonic saline nebulization in patients with cystic fibrosis exacerbation. The study assesses whether these devices facilitate the easier evacuation of retained secretions, shorten bronchial drainage time, and improve pulmonary function test results. Participants are randomly assigned to specific groups (Group I - inhalation with O-PEP, Group II - inhalation with PEP, Group III - control group, standard inhalation) using a calendar formula (day of the month divided by 3). Each group performs bronchial drainage following the same protocol: autogenic drainage and a device with positive variable expiratory pressure (device name: Pari O-PEP).

The main questions the study aims to answer are: 1. Does implementing inhalation devices improve functional test indicators and the amount of mucus expectorated during inhalation? 2. Are there differences in effectiveness between the groups?

ELIGIBILITY:
Inclusion Criteria:

* written consent of the patient and/or guardian,
* no disease complications (within the last 2 months) in the form of: active haemoptysis, chest surgeries, surgical procedures in the area of the esophagus (esophageal varices), otitis media,
* Age above 10 years,
* the ability to perform correctly lung function tests and FEV1 value above 20% predicted,
* the presence of respiratory symptoms indicating exacerbation of the disease, i.e. increasing of cough, increasing of dyspnoea, decrease in FEV1 by 10% or more from a previously recorded value.

Exclusion Criteria:

* Lack of written consent for the study
* Hemoptysis within the last 2 months
* History of pneumothorax
* Current otitis media
* Age below 10 years
* FEV1 value below 20% of the predicted value
* Surgical procedures in the area of the oesophagus (esophageal varices)
* Intolerance to the PEP or O-PEP device

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Pulmonary Function Test (PFT) | From baseline to study completion, the average duration is 10 days.
  Measured indicators: Bodyplethysmographie: FEV1, FVC, volume measurement (L). Change from baseline during hospitalization (at least 8 days).
1. Pulmonary Function Test (PFT) | From baseline to study completion, the average duration is 10 days.
  Measured indicators: Bodyplethysmographie: MEF 50, flow measurement (l/s). Change from baseline during hospitalization (at least 8 days).
1.2 Pulmonary Function Test (PFT) | From baseline to study completion, the average duration is 10 days.
  Measured indicators: Impulse Oscillometry, IOS: R20, R5 kilopaskal per litre per second (kPa/l/s). Change from baseline during hospitalization (at least 8 days).
Survey Cystic Fibrosis Questionnaire-Revised (CFQ-R) | From baseline to study completion, the average duration is 10 days.
  A survey assessing the quality of life, dedicated to people with cystic fibrosis. The survey includes questions on: physical, vitality, emotion, eat, treatment burden, health perception, social, body, role, weight, respiratory, digestion. The survey is intended for people with cystic fibrosis and their parents from 6 years of age. Interpretion: a score scale scale title: Manual scoring for the Cystic Fibrosis Questionnaire-Revised (CFQ-R), Teen/adult: Minimum values 1 Maximum values 196, Parents: Minimum values 1 Maximum values 157, Child 12 to 13: minumum values 1 maximum values 128, Child 6 to 11: minumum values 1 maximum values 128.

OTHER OUTCOMES:
Sputum expectorated. | From baseline to study completion, the average duration is 10 days.
  Volume measurement [ml], during inhalation and during physiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Warzeszak, Principal Investigator — National Tuberculosis and Lung Diseases Research Institute
Locations (2):
- Poland (2):
  - National Tuberculosis and Lung Diseases Research Institute, Rabka-Zdrój, Malopolska
  - National Institute Tuberculosis and Lung Diesases, Rabka-Zdrój, Małopolska

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murray MP, Pentland JL, Turnbull K, MacQuarrie S, Hill AT. Sputum colour: a useful clinical tool in non-cystic fibrosis bronchiectasis. Eur Respir J. 2009 Aug;34(2):361-4. doi: 10.1183/09031936.00163208. PMID 19648517
- [Background] San Miguel-Pagola M, Reychler G, Cebria I Iranzo MA, Gomez-Romero M, Diaz-Gutierrez F, Herrero-Cortina B. Impact of hypertonic saline nebulisation combined with oscillatory positive expiratory pressure on sputum expectoration and related symptoms in cystic fibrosis: a randomised crossover trial. Physiotherapy. 2020 Jun;107:243-251. doi: 10.1016/j.physio.2019.11.001. Epub 2019 Nov 11. PMID 32026826
- [Background] Orlik T, Sands D. Application of positive expiratory pressure *PEP* in cystic fibrosis patient inhalations. Dev Period Med. 2015 Jan-Mar;19(1):50-9. PMID 26003070
- [Background] Berlinski A. In vitro evaluation of positive expiratory pressure devices attached to nebulizers. Respir Care. 2014 Feb;59(2):216-22. doi: 10.4187/respcare.02698. Epub 2013 Aug 6. PMID 23920213
- [Background] Chatham K, Ionescu AA, Nixon LS, Shale DJ. A short-term comparison of two methods of sputum expectoration in cystic fibrosis. Eur Respir J. 2004 Mar;23(3):435-9. doi: 10.1183/09031936.04.00084904. PMID 15065835